CLINICAL TRIAL: NCT03495765
Title: An Open-label, Multi-centre, 12-month Study to Evaluate the Comparative Efficacy of Lucentis (Ranibizumab) 0.5mg Intravitreal Injection in Patients With Diabetic Macular Oedema (DME) With Well Controlled and Poorly Controlled Diabetes Mellitus ('CONTROL' Study)
Brief Title: To Evaluate the Comparative Efficacy of Lucentis (Ranibizumab) 0.5mg Intravitreal Injection in Patients With Diabetic Macular Oedema (DME) With Well Controlled and Poorly Controlled Diabetes Mellitus
Acronym: CONTROL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marsden Eye Specialists (Other)
Responsible Party: Principal Investigator, Dr Jennifer Arnold, Principal Investigator, Marsden Eye Specialists
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Control1
Record Dates: First submitted 2018-04-03; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Macular Oedema
Keywords: Diabetic macular oedema; Lucentis
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Well controlled (Active Comparator): Eligibile people with diabetic macular oedema and HBA1C < 7.5
  Interventions: Drug: Ranibizumab
- Poorly controlled (Active Comparator): eligible people with Diabetic macular oedema and HBAIC >10.0
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5mcg via intravitreal injection to study eye up to monthly
  Other Names: Lucentis

SUMMARY:
To demonstrate the comparative effectiveness of 12 months of Lucentis (ranibizumab) in patients with well controlled compared to those with poorly controlled diabetes using an PRN treatment schedule.

DETAILED DESCRIPTION:
To demonstrate the comparative effectiveness of Lucentis (ranibizumab) in patients with well controlled compared to those with poorly controlled diabetes.

The primary endpoint for the study will be the mean change in best-corrected visual acuity (BCVA) from baseline to Month 12.

Two groups of patients, based on HbA1c levels will be entered into the trial -

1. patients with a recent HbA1c level < 7.5 % (the 'well controlled' subgroup) and
2. patients with a recent HbA1c level ≥ 10.0% (the 'poorly controlled' subgroup).

Ranibizumab treatment will be administered over the 12-month period, initial 3 monthly injections, followed by 'as needed' protocol using the following principles:

Monthly ranibizumab injections would be suspended when:

* No further BCVA improvement from treatment at the last 2 consecutive follow up visits OR
* BCVA letter score >84 (6/6) at the last 2 consecutive follow up visits

Monthly ranibizumab injections would be reinitiated when:

• Decrease in BCVA due to DME progression in the opinion of the investigator Laser treatment could also be administered from 3 months after study initiation, according to the investigators decision, in accordance with ETDRS guidelines, and at intervals of at least 3 months from the last treatment.

Visit schedule: Screening visit then monthly visits for 12 visits (total of 13 visits)

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with diabetes > 21 years of age who have signed an informed consent
* Patients with either Type 1 or Type 2 diabetes mellitus (according to ADA or WHO guidelines) with HbA1c levels either < 7.5% or ≥ 10.0% at screening (visit 1) as measured within the last 3 months.
* Patients with visual impairment due to either focal or diffuse DME in at least one eye who are eligible for laser treatment in the opinion of the investigator. The study eye must fulfill the following criteria at Visit 1 (if both eyes are eligible, the study eye will be selected by the investigator, based on potential for improvement): i) BCVA score between 73 and 39 letters, inclusively, using LogMAR visual acuity testing charts at 4 metres (or at the equivalent appropriate testing distance for the chart size) (approximate Snellen equivalent between 6/12 (20/40) and 6/48 (20/160); ii) the decrease in vision is due to DME but not due to other causes, in the opinion of the investigator
* OCT foveal centre point thickness ≥ 350µm on Spectral Domain OCT (≥300 µm on Time domain OCT / STRATUS)
* Medication for the management of diabetes should have been stable within the 3 months prior to randomisation

Exclusion Criteria:

* Concomitant conditions in the study eye which could, in the opinion of the investigator, prevent the improvement of visual acuity on study treatment
* Active intraocular inflammation (grade trace or above) in either eye
* Any active infection (e.g. conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in either eye
* History of uveitis in either eye
* Structural damage within 1 disc diameter of the center of the macula in the study eye likely to preclude an improvement in visual acuity following the resolution of macular oedema, including (geographic) atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), or organized hard exudates plaques
* Ocular disorders in the study eye that may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the 12-month study period, including retinal vascular occlusion, retinal detachment, epiretinal membrane, macular hole, or choroidal neovascularization of any cause (e.g., AMD, ocular histoplasmosis, or pathologic myopia)
* Uncontrolled glaucoma in the study eye (according to investigator's judgment)
* Neovascularization of the iris in study eye
* Evidence of vitreomacular traction in study eye, shown either clinically or on OCT
* Panretinal laser photocoagulation in the study eye within 6 months (in order to exclude patients with active proliferative disease) or focal/grid laser photocoagulation in the study eye within 3 months prior to study entry
* Treatment with anti-angiogenic drugs: pegaptanib sodium, anecortave acetate, bevacizumab, ranibizumab, aflibercept (VEGF-Trap) within 3 months to study eye
* Intravitreal corticosteroids in either eye within 6 months prior to randomisation
* Any intraocular surgery in the study eye within 3 months prior to randomisation
* History of vitrectomy in study eye
* Phakic study eye with a history of intravitreal corticosteroid treatment (due to the likely late increase in secondary cataract)
* Ocular conditions in the study eye that is likely to require chronic concomitant therapy with topical ocular or systemically administered corticosteroids
* History of disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that might affect the interpretation of the results of the study, or that would renders the patient at high risk from treatment complications
* Renal failure requiring dialysis or renal transplant OR renal insufficiency with creatinine levels >2.0 mg/dl
* Untreated diabetes mellitus
* Severe (blood pressure systolic > 160 mmHg OR diastolic > 100 mmHg)
* Current use of or likely need for systemic medications known to be toxic to the lens, retina or optic nerve, including Deferoxamine, Chloroquine/ hydroxychloroquine (Plaquenil), Tamoxifen, Phenothiazines and Ethambutol
* Known hypersensitivity to ranibizumab or any component of the ranibizumab formulation
* Previous participation in any clinical studies of investigational drugs (excluding vitamins and minerals) within 1 month (or a period corresponding to 5 half-lives of the investigational drug, whatever is longer) prior to randomisation
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Pregnant or nursing (lactating) women.
* Inability to comply with study or follow-up procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for the study will be the mean change in best-corrected visual acuity (BCVA) from baseline to the mean level at Month 12. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Marsden Eye Specialists, Paramatta, New South Wales, Australia